CLINICAL TRIAL: NCT02472782
Title: Prospective,Non-interventional Study Investigating Possible Correlation Between Adherence to Postmenopausal and Steroid Induced Osteoporosis Treatment and Physicians' Perception Regarding Osteoporosis Medication
Brief Title: Adherence to Osteoporosis Treatment and Physicians' Perception Regarding Osteoporosis Medication
Acronym: IASIS
Status: Completed | Type: Observational
Sponsor: 251 Hellenic Air Force & VA General Hospital (Other)
Collaborators: Hellenic Osteoporosis Foundation (www.http://heliost.gr/en/) (Unknown)
Responsible Party: Principal Investigator, Dr Polyzois Makras, Deputy Director, Dpt of Endocrinology & Diabetes, 251 Hellenic Air Force & VA General Hospital
Other Study IDs: 076/AD7592/S1684/6-5-2015
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis, Steroid Induced
Keywords: osteoporosis; quality of life; adherence; treatment
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Teriparatide — The study will include patients from pre-defined groups of individuals (postmenopausal, male, and steroid-induced osteoporosis) who would any way receive teriparatide for their condition according to standard medical practice and Greek treatment guidelines
  Other Names: osteo-anabolic treatment

SUMMARY:
This is a study aiming to investigate a possible correlation between the parameters affecting the physicians' therapeutic choice with the patients' overall adherence to osteoporosis treatment. Secondary end-points include correlation between the parameters affecting the physicians' therapeutic choice and the patients' quality of life as well as the evaluation of the whole osteoporosis treatment approach of orthopedic surgeons in Greece (diagnostic means, use of diagnostic and treatment guidelines, methodology of follow - up).

DETAILED DESCRIPTION:
The study will include 100 orthopedic surgeons from the private sector working in private offices. The selection of this group of physicians resides on the fact that orthopedic surgeons working in private offices hold more than 60% of osteoporosis prescriptions in Greece.

Each physician will fill once a questionnaire regarding the parameters affecting his/her choice of osteoporosis treatment before entering any patient in the study. Following the completion of the questionnaire every physician will recruit up to 10 patients in the study who are eligible for osteoanabolic treatment (teriparatide) according to standard medical practice and the Greek osteoporosis treatment guidelines.

Each patient will receive teriparatide up to 24 months while he/she will fill the Greek EQ5D questionnaire on months: 0,12,24 or at early discontinuation. Adherence to treatment will be evaluated at the same time points as well as on monthly telephone interviews.

Both the adherence to treatment and the possible alteration of patients' quality of life (evaluated through the EQ5D questionnaire) during the study will be correlated with the parameters affecting the initial therapeutic decision of the physician

ELIGIBILITY:
Inclusion Criteria:

* Female patients with postmenopausal osteoporosis (T-score ≤-2,5 SD at any skeletal site) under osteoporosis treatment (except teriparatide) for at least one year with a history of ≥ low-energy fracture during the last 10 years prior the study.
* Male patients ≥ 50 years old with idiopathic osteoporosis (T-score ≤-2,5 SD at any skeletal site) under osteoporosis treatment (except teriparatide) for at least one year with a history of ≥ low-energy fracture during the last 10 years prior the study.
* Male and female patients with steroid-induced osteoporosis (T-score ≤-2,5 SD at any skeletal site) under osteoporosis treatment (except teriparatide) for at least one year with a history of ≥ low-energy fracture during the last 10 years prior the study.

Exclusion Criteria:

* Prior use of teriparatide or PTH(1-84)
* Hypersensitivity to teriparatide regimen.
* Pregnancy and lactation.
* Hypercalcamia.
* Renal deficiency (eGFR < 30 ml/min).
* Other bone metabolic diseases (including hyperparathyroidism and Paget's disease) except primary osteoporosis or steroid induced osteoporosis .
* Uninterpretable increases of alkaline phosphatase (ALP)
* Prior skeletal radiotherapy.
* Skeletal malignancies or bone metastases

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with postmenopausal osteoporosis
  Male patients ≥ 50 years old with idiopathic osteoporosis
  Male and female patients with steroid-induced osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 851 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Adherence to osteoporosis treatment assessed by medication possession ratio (MPR) | 2 years
  Adherence to osteoporosis treatment assessed by medication possession ratio Adherence to osteoporosis treatment assessed by medication possession ratio (MPR) and correlation with the parameters affecting the physicians' therapeutic choices

SECONDARY OUTCOMES:
Quality of life assessed by EQ5D questionnaire | 2 years
  Quality of life assessed by EQ5D questionnaire and correlation with the parameters affecting the physicians' therapeutic choice

CONTACTS AND LOCATIONS:
Overall Officials: George Lyritis, Professor, Study Chair — Hellenic Osteoporosis Foundation
Locations (1):
- 251 Hellenic Air Force & VA General Hospital, Athens, Attica, Greece

REFERENCES:
- [Background] Briot K, Ravaud P, Dargent-Molina P, Zylberman M, Liu-Leage S, Roux C. Persistence with teriparatide in postmenopausal osteoporosis; impact of a patient education and follow-up program: the French experience. Osteoporos Int. 2009 Apr;20(4):625-30. doi: 10.1007/s00198-008-0698-8. Epub 2008 Jul 26. PMID 18661089
- [Background] Lyritis GP, Rizou S, Galanos A, Makras P. Incidence of hip fractures in Greece during a 30-year period: 1977-2007. Osteoporos Int. 2013 May;24(5):1579-85. doi: 10.1007/s00198-012-2154-z. Epub 2012 Oct 13. PMID 23064370
- [Background] Cramer JA, Roy A, Burrell A, Fairchild CJ, Fuldeore MJ, Ollendorf DA, Wong PK. Medication compliance and persistence: terminology and definitions. Value Health. 2008 Jan-Feb;11(1):44-7. doi: 10.1111/j.1524-4733.2007.00213.x. PMID 18237359
- [Background] Huybrechts KF, Ishak KJ, Caro JJ. Assessment of compliance with osteoporosis treatment and its consequences in a managed care population. Bone. 2006 Jun;38(6):922-8. doi: 10.1016/j.bone.2005.10.022. Epub 2005 Dec 5. PMID 16330270
- [Background] Hadji P, Claus V, Ziller V, Intorcia M, Kostev K, Steinle T. GRAND: the German retrospective cohort analysis on compliance and persistence and the associated risk of fractures in osteoporotic women treated with oral bisphosphonates. Osteoporos Int. 2012 Jan;23(1):223-31. doi: 10.1007/s00198-011-1535-z. Epub 2011 Feb 10. PMID 21308365
- [Background] Netelenbos JC, Geusens PP, Ypma G, Buijs SJ. Adherence and profile of non-persistence in patients treated for osteoporosis--a large-scale, long-term retrospective study in The Netherlands. Osteoporos Int. 2011 May;22(5):1537-46. doi: 10.1007/s00198-010-1372-5. Epub 2010 Sep 14. PMID 20838773
- [Background] Arden NK, Earl S, Fisher DJ, Cooper C, Carruthers S, Goater M. Persistence with teriparatide in patients with osteoporosis: the UK experience. Osteoporos Int. 2006;17(11):1626-9. doi: 10.1007/s00198-006-0171-5. Epub 2006 Jul 6. PMID 16823543